CLINICAL TRIAL: NCT02485522
Title: Diet and Stool Metabolites in Women With Fecal Incontinence
Brief Title: Diet and Stool Metabolites in Fecal Incontinence
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 822653
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; diet; nutrition; metabolites; stool; FI
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Fecal incontinence: Women age >18 years old with a diagnosis of fecal incontinence
  Interventions: Other: No Intervention
- Controls: Women age >18 without a diangosis of fecal incontinence
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
Fecal Incontinence (FI) is a debilitating and common condition with a prevalence ranging from 7-15% in community dwelling women. FI has an immense impact on quality of life and is associated with increased care giver burden, increased rates of institutionalization, and significant cost burden in older women. Traditionally believed to be primarily caused by child birth injury, recent studies show that the typical age of onset of FI is age 40 which is remote from child birth. Treatment options for FI are limited because the mechanism underlying FI in older women are poorly understood. The overriding goal of this project is to investigate the relationship between diet, stool metabolites and fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18,
* parous women with fecal incontinence (defined as any uncontrolled loss of liquid or solid fecal material that occurs at least monthly over the last 3 months that is bothersome enough to desire treatment),
* current negative colon cancer screening

Exclusion Criteria:

* Current bloody diarrhea,
* current or past diagnosis of colorectal or anal malignancy,
* diagnosis of inflammatory bowel disease,
* recent antibiotic treatment,
* history of immune deficiency diseases,
* history of recent treatment with immune suppressant medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with fecal incontinence from an outpatient GYN clinic.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Stool butyrate levels | within 1 week of collection
Pattern of dietary intake by indicator | 1 year

SECONDARY OUTCOMES:
Stool levels of global metabolites | within 1 week of collection

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States